CLINICAL TRIAL: NCT04539678
Title: Retrospective and Prospective Multicenter Study Evaluating the Impact of Treatment With Cytoreducing Agents on the Recurrence of Thrombosis in Thrombotic Patients With a Diagnosis of Myeloproliferative Neoplasia and Normal Blood Counts - a FIM Study
Brief Title: SYTHROM Cohort, Myeloproliferative Neoplasia With Normal CBC and Thrombotic Complications
Acronym: SYTHROM
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: French Intergroup of Myeloproliferative syndromes (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC20_0141
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Thrombotic Patients; Diagnosis of Myeloproliferative Neoplasia; Impact of Treatment With Cytoreducing Agent
Keywords: Thrombosis; Myeloproliferative neoplasm; Hydroxyurea; Interferon
MeSH Terms: conditions — Thrombosis; Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Among the etiologies of thrombosis, myeloproliferative neoplasia (MPN) is quite rare but should be investigated in case of thrombosis of atypical localization (digestive or cerebral) or in the context of recurrent idiopathic thrombosis in a young subject. Thrombosis could reveal an underlying MPN through the identification of a JAK2 V617F mutation. Rarely, MPN with thrombotic complications present with normal complete blood count(CBC). In case of a MPN with a thrombotic event but without CBC abnormality, anti-thrombotic treatment is recommended. But there is no recommendation for the indication of cytoreductive therapy and the clinician's decision is often empirical.

One of the major complications of for essential thrombocythemia (ET) or polycythemia vera (PV) is thrombosis and an age over 60 is a major risk factor. The treatment of thrombosis associated with TE or PV is based on recommendations the main therapeutic objective of which is to reduce the thrombotic risk. The combination of a cytoreducing agent and antithrombotic treatment is thus proposed in high-risk patients. The efficacy of this management is monitored by assessing CBC with the objective of normalization at <400 G/L of platelets for ET patients and <45% hematocrit in case of PV.

The absence of abnormal CBC makes it difficult to justify cytoreduction. The benefit of such a therapy in this context has not been clinically demonstrated. If a cytoreductive therapy is initiated, no biological parameters are available to assess the response to treatment.

The objective of this observational study is to evaluate the incidence of recurrence of thrombosis in patients whose thrombotic event revealed an underlying MPN with normal CBC. A comparison of groups treated or not with cytoreductive agents will be performed. Longitudinal monitoring of the patients will provide a better understanding of the nature and kinetics of hematological changes in these patients.

DETAILED DESCRIPTION:
This study is observational and multicentric.In a first part, patients will be retrospectively included. Baseline clinical and biological data obtainedat the time of MPN diagnosis of MPN with normal CBC following venous or arterial thrombosis will be recorded and follow-up data will be collected in an e-CRF. In a second part, patients will be included prospectively and diagnostic and follow-up data will be collected. Whether or not to initiate treatment with a cytoreduction treatment is left to the discretion of the clinician.

ELIGIBILITY:
Inclusion Criteria :

* Adult ≥18 years old
* Diagnosis of a deep arterial or venous thrombotic event verified by imaging (Doppler or CT scan)
* Diagnosis of MPN with normal CBC according to WHO 2017 criteria characterized by the detection of a molecular abnormality JAK2V617F mutation (regardless of allelic load), CALR or MPL and/or a bone marrow biopsy with abnormalities in favor of MPN.
* Normal blood cell count not suggestive of polycythemia vera (hematocrit<48% and hemoglobin<16g/dL for women; hematocrit<49% and hemoglobin<16.5g/dL for men), essential thrombocythemia (platelets<450 G/L) nor myelofibrosis (white blood cell count<11 G/L, no anemia or erythromyelemia associated with splenomegaly) at the time of the thrombotic event.

Exclusion Criteria :

* Minors (<18 years of age)
* Microcirculation disorders (erythromelalgia, headaches, paresthesia, ischemia of the extremities)
* Superficial or deep arterial or venous thrombosis NOT verified by imaging
* Diagnosis or history of TE, PV or myelofibrosis at time of first thrombotic event
* Diagnosis of mixed myelodysplastic/myeloproliferative syndrome
* Diagnosis of unclassifiable MPN with excess blasts at the onset or signs of myelodysplasia as defined by the WHO 2017 classification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thrombosis recurrence :treated and untreated patients with cytoreductive agents
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of recurrence of thromboembolic events after the initial thrombosis leading to the diagnosis of MPN | 24 months follow-up
  The diagnosis of thromboembolic events must be confirmed by imaging

SECONDARY OUTCOMES:
Cumulative incidence of hematological progression to essential thrombocythemia, polycythemia vera, secondary myelofibrosis or acute transformation | 24 months follow-up
  Hematological progression criteria will be based on the WHO classification
Cumulative incidence of recurrence of thromboembolic events according to the type and duration of anticoagulant or anti-aggregant treatment | 24 months follow-up
  The diagnosis of thromboembolic event must be confirmed by imaging

CONTACTS AND LOCATIONS:
Overall Officials: Yannick LE BRIS, PhD, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kiladjian JJ, Cervantes F, Leebeek FW, Marzac C, Cassinat B, Chevret S, Cazals-Hatem D, Plessier A, Garcia-Pagan JC, Darwish Murad S, Raffa S, Janssen HL, Gardin C, Cereja S, Tonetti C, Giraudier S, Condat B, Casadevall N, Fenaux P, Valla DC. The impact of JAK2 and MPL mutations on diagnosis and prognosis of splanchnic vein thrombosis: a report on 241 cases. Blood. 2008 May 15;111(10):4922-9. doi: 10.1182/blood-2007-11-125328. Epub 2008 Feb 4. PMID 18250227
- [Background] De Stefano V, Fiorini A, Rossi E, Za T, Farina G, Chiusolo P, Sica S, Leone G. Incidence of the JAK2 V617F mutation among patients with splanchnic or cerebral venous thrombosis and without overt chronic myeloproliferative disorders. J Thromb Haemost. 2007 Apr;5(4):708-14. doi: 10.1111/j.1538-7836.2007.02424.x. Epub 2007 Jan 29. PMID 17263783
- [Background] Levraut M, Legros L, Drappier C, Bene MC, Queyrel V, Raynaud S, Martis N. Low prevalence of JAK2 V617F mutation in patients with thrombosis and normal blood counts: a retrospective impact study. J Thromb Thrombolysis. 2020 Nov;50(4):995-1003. doi: 10.1007/s11239-020-02100-z. PMID 32266587
- [Background] Barbui T, Thiele J, Passamonti F, Rumi E, Boveri E, Ruggeri M, Rodeghiero F, d'Amore ES, Randi ML, Bertozzi I, Marino F, Vannucchi AM, Antonioli E, Carrai V, Gisslinger H, Buxhofer-Ausch V, Mullauer L, Carobbio A, Gianatti A, Gangat N, Hanson CA, Tefferi A. Survival and disease progression in essential thrombocythemia are significantly influenced by accurate morphologic diagnosis: an international study. J Clin Oncol. 2011 Aug 10;29(23):3179-84. doi: 10.1200/JCO.2010.34.5298. Epub 2011 Jul 11. PMID 21747083
- [Background] Barbui T, Finazzi G, Carobbio A, Thiele J, Passamonti F, Rumi E, Ruggeri M, Rodeghiero F, Randi ML, Bertozzi I, Gisslinger H, Buxhofer-Ausch V, De Stefano V, Betti S, Rambaldi A, Vannucchi AM, Tefferi A. Development and validation of an International Prognostic Score of thrombosis in World Health Organization-essential thrombocythemia (IPSET-thrombosis). Blood. 2012 Dec 20;120(26):5128-33; quiz 5252. doi: 10.1182/blood-2012-07-444067. Epub 2012 Oct 1. PMID 23033268
- [Background] Pearson TC, Wetherley-Mein G. Vascular occlusive episodes and venous haematocrit in primary proliferative polycythaemia. Lancet. 1978 Dec 9;2(8102):1219-22. doi: 10.1016/s0140-6736(78)92098-6. PMID 82733
- [Background] Barosi G, Birgegard G, Finazzi G, Griesshammer M, Harrison C, Hasselbalch HC, Kiladjian JJ, Lengfelder E, McMullin MF, Passamonti F, Reilly JT, Vannucchi AM, Barbui T. Response criteria for essential thrombocythemia and polycythemia vera: result of a European LeukemiaNet consensus conference. Blood. 2009 May 14;113(20):4829-33. doi: 10.1182/blood-2008-09-176818. Epub 2009 Mar 10. PMID 19278953